CLINICAL TRIAL: NCT00360438
Title: Pharmacokinetic Evaluation of Rasburicase Dosed for 5 Consecutive Days as Uricolytic Therapy in Adult Patients With Leukemia and/or Lymphoma at High or Potential Risk of Tumor Lysis Syndrome (TLS)
Brief Title: Pharmacokinetic Evaluation of Rasburicase in Patients With Leukemia and/or Lymphoma at High Risk of TLS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-0298
Record Dates: First submitted 2006-08-02; First posted 2006-08-04 (Estimated); Last update posted 2012-08-01 (Estimated); Status verified 2012-07

CONDITIONS: Leukemia; Lymphoma; Tumor Lysis Syndrome
Keywords: Leukemia; Lymphoma; Tumor Lysis Syndrome; TLS; Rasburicase; Elitek
MeSH Terms: conditions — Leukemia; Lymphoma; Tumor Lysis Syndrome | interventions — rasburicase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rasburicase (Experimental)
  Interventions: Drug: Rasburicase

INTERVENTIONS:
Drug: Rasburicase — 0.15mg/kg intravenously over 30 minutes once per day for 5 consecutive days.
  Other Names: Elitek

SUMMARY:
Primary

1. To determine the pharmacokinetic (PK) parameters of rasburicase in adult patients with leukemia and/or lymphoma at high risk or potential risk of tumor lysis syndrome (TLS)

Secondary

1. To evaluate plasma uric acid AUC from baseline (within 4 hours prior to first rasburicase treatment) through 48 hours after the last per-protocol planned administration of rasburicase treatment;
2. To evaluate the safety of rasburicase in adult patients with leukemia and/or lymphoma.
3. To evaluate incidence, duration, and type of immune responses (IgG, IgE, and neutralizing antibody) to rasburicase.

DETAILED DESCRIPTION:
Rasburicase is designed to help decrease or prevent the high level of uric acid that may occur during the start of chemotherapy. A high level of uric acid may lead to reduced kidney function or kidney failure.

TLS occurs when high uric acid levels are caused by breakdown of tumor cells after the start of chemotherapy. The dead tumor cells can release uric acid and other symptoms of kidney failure, such as excessive amounts of potassium and phosphorus, into the blood.

Before you can start treatment on this study, you will have "screening tests." These tests will help the doctor decide if you are eligible to take part in this study. Your complete medical history will be recorded, and you will have a physical exam, including measurement of your vital signs (blood pressure, heart rate, temperature, and breathing rate), height, and weight. You will have blood drawn (about 2 tablespoons) for routine tests. Women who are able to have children must have a negative blood (a sample will be used from the routine blood draw) or urine pregnancy test.

If you are found to be eligible to take part in this study, you will receive rasburicase by a needle in your vein over 30 minutes once a day for 5 days in a row. You will receive chemotherapy within 4-24 hours after your first dose of rasburicase.

On Days 1-5 (study drug treatment period), you will have a physical exam, including measurement of your vital signs. During this time, you will have blood drawn (about 2 tablespoons each) once a day for routine tests.

You will have blood drawn (less than 1 teaspoon each) for PK testing at different time points throughout this study. PK tests measure the level of the study drug in the blood at different times. You will have a total of 14 samples drawn. Your blood will be drawn on Day 1 before your dose of rasburicase and then at 30 minutes and at 4, 8, 24, 48, 72, 96, 96.5,100,104,120 (Day 6),168 (Day 8), and 336 (Day 15) hours after your dose of the study drug.

You will have blood drawn (less than 1 teaspoon each) to measure the level of uric acid in your blood at different time points throughout this study so that researchers can learn the effectiveness of the study drug on your disease. You will have a total of 7 samples drawn. Your blood will be drawn on Day 1 before your dose of rasburicase and then at 4, 24, 48, 72, 96,120 (Day 6), and 144 (Day 7) hours after your dose of the study drug.

You will also have blood drawn (less than 1 teaspoon each) for antibody testing at different time points throughout this study. Antibody testing is a method to check for proteins (IgG) made by your body that show that your body is reacting to rasburicase. You will have at least 5 samples drawn. Your blood will be drawn on Day 1 before your dose of rasburicase and then on Day 14, Day 35, and at 3 and 6 months after your dose of the study drug.

If you have a positive IgG (antibody protein) at the 6-month blood draw for antibody testing, you will continue to have blood drawn (less than 1 teaspoon) every 6 months until your antibody protein is negative.

If you experience any side effects related to allergic reactions during treatment with the study drug (up to 30 days after your last dose of the study drug), you will have an additional blood draw (less than 1 teaspoon) for antibody testing within 48 hours after having the reaction.

You will be taken off this study if your disease gets worse or you experience any intolerable side effects.

You will have assessments after the end of your study drug treatment (from Days 1 to 5). These assessments will include a physical exam, including measurement of your vital signs, on Days 14 and 35. You will also have blood drawn (about 2 tablespoons each) for routine tests on Days 8 and 14.

This is an investigational study. Rasburicase is authorized by the FDA for use (in adults) in research only. Rasburicase will be provided free of charge during this study. Up to 20 patients will take part in this multicenter study. Up to 20 can be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Age >/= 18
2. Risk of TLS: A. High risk: hyperuricemia of malignancy; diagnosis of aggressive lymphoma/leukemia based on Revised European-American Lymphoma (REAL) classification; acute myeloid leukemia in blast crisis; high grade myelodysplastic syndrome only if they have >10% bone marrow blast involvement and given aggressive treatment similar to AML; OR B. Potential risk: diagnosis of aggressive lymphoma/leukemia based on (REAL) classification. Plus one or more of the following criteria: LDH >/=2 x ULN; Stage III-IV disease; Stage I-II disease with at least 1 lymph node/tumor >5cm in diameter.
3. ECOG performance status 0-3
4. Life expectancy >3 months
5. Negative pregnancy test (females of child bearing potential) within </=2 weeks of rasburicase dose and use of efficient contraceptive method (both males and females). Pregnancy test may be performed on serum (HCG) or urine (HCG)
6. Signed written informed consent (approved by the Institutional Review Board/Ethics Committee) obtained prior to study entry

Exclusion Criteria:

1. Patient receiving any investigational drug for hyperuricemia within 30 days of planned first treatment with rasburicase
2. Pregnancy or lactation
3. Known history of significant allergy problem or documented history of asthma or asthmatic bronchitis
4. Known history of glucose-6-phosphate dehydrogenase deficiency
5. Known history of hemolysis and methemoglobinemia
6. Positive tests for HBs antigen, HCV antibodies, or HIV-1, 2 antibodies
7. Hypersensitivity to uricases or any of the excipients
8. Previous therapy with urate oxidase
9. Other conditions unsuitable for participation in the trial in the Investigator's opinion
10. Unwilling to comply with the requirements of the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2006-07; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Effectiveness of rasburicase in treatment of patients with leukemia and/or lymphoma who are at high or potential risk for TLS. | 4 Years

CONTACTS AND LOCATIONS:
Overall Officials: Saroj Vadhan-Raj, M.D., Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org